CLINICAL TRIAL: NCT06037408
Title: The Effect of Sodium Pyruvate Nasal Spray on Coughing in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: The Effect of N115 on Coughing in IPF Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cellular Sciences, inc. (Industry)
Collaborators: Family First Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00072822
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20mM sodium pyruvate nasal spray treatment (Experimental)
  Interventions: Drug: 20mM sodium pyruvate nasal spray
- Saline placebo control (Placebo Comparator)
  Interventions: Other: Saline Placebo control nasal spray

INTERVENTIONS:
Drug: 20mM sodium pyruvate nasal spray — The product is a 20 mM (0.2%, 2.2 mg/mL) sodium pyruvate nasal spray in 0.9% sodium chloride with benzalkonium chloride preservative, pH 7.2 (N115). Subjects will self-administer 3 squirts per nostril of the nasal spray, 3 times daily; upon wakening, noon/midday, and before bedtime.
  Arms: 20mM sodium pyruvate nasal spray treatment
Other: Saline Placebo control nasal spray — The placebo is 0.9% sodium chloride with benzalkonium chloride preservative, pH 7.2. Subjects will self-administer 3 squirts per nostril of the nasal spray, 3 times daily; upon wakening, noon/midday, and before bedtime.
  Arms: Saline placebo control

SUMMARY:
The purpose of this clinical trial is to administer a sodium pyruvate nasal spray that eliminates nasal oxidative stresses, caused by oxygen radicals, and demonstrate the efficacy of sodium pyruvate to reduce coughing and increase lung functions in patients with idiopathic pulmonary fibrosis. This will be a 21-day double-blinded randomized placebo-controlled trial designed to determine if patients with idiopathic pulmonary fibrosis treated with 20mM sodium pyruvate in 0.9% sodium chloride nasal spray solution will have reduced chronic coughing, as well as increased lung function (FEV1, FVC endpoints of 12% or more within the first week) and improved FEV1/FVC ratios.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) belongs to a group of conditions called interstitial lung diseases (also known as ILD), which describes lung diseases that involve inflammation or scarring in the lung. IPF is a chronic progressive lung disorder associated with excessive tissue remodeling, scarring, and fibrosis, which makes the lungs unable to effectively transport oxygen into the bloodstream resulting in decreased lung function and increased nasal inflammation with increased mucus and coughing and poor quality of life. IPF usually affects people between the ages of 30 and 70. The most common signs and symptoms of IPF are shortness of breath and persistent dry, hacking cough. Many affected individuals also experience a loss of appetite and gradual weight loss. Most affected individuals survive 3 to 5 years after their diagnosis. However, the course of the disease is highly variable; some affected people become seriously ill within a few months, while others may live with the disease for a decade or longer. In most cases, IPF is sporadic and results from environmental damage to the lungs and not genetic factors. However, a small percentage of people have genetic risk factors resulting in familial pulmonary fibrosis.

Sodium pyruvate is a natural antioxidant of the human body and as an antioxidant it has been shown to significantly reduce inflammatory agents throughout the human body, including the lungs and nasal passages, allowing nasal nitric oxide to reach the lungs to increase bronchodilation. In addition to 8 human clinical studies conducted on the effect of inhaled sodium pyruvate on the lungs, 7 human nasal inhalation clinical studies were conducted using a sodium pyruvate nasal spray which showed decreased nasal inflammation, a reduction in inflammatory cytokines, and when measured, demonstrated an increase in lung functions, a decrease in coughing, including in patients with pulmonary fibrosis and IPF. Cellular Sciences received Orphan Drug designations for Cystic Fibrosis and Interstitial lung Disease.

A previous open label phase 2, 21-day, sub-chronic clinical trial was conducted that included 15 patients with pulmonary fibrosis (9 with pulmonary fibrosis and chronic obstructive pulmonary disease (COPD) and 6 with idiopathic pulmonary fibrosis without COPD) that remained on their normal medications but were also administered a 20 mM (2.2 mg/mL) sodium pyruvate nasal spray 3 times per day for 22 days. The data from this study showed that coughing episodes per 24 hours, and especially at night, were significantly reduced in all 15 patients on day 8 by 30% (p = 0.007) and continued to decrease on day 14 by 55% (p = 0.0001) and on the 22 day of the trial, coughing decreased by 59% (p = 0.0001). This correlated with a significant (p = 0.010) improvement in nasal irritation/erythema with most patients being free of irritation by day 22 (p < 0.001); and a significant (p = 0.010) increase in the group average expelled NO by day 8. A significant (p = 0.010) improvement in lung function (breathing) was observed in all patients with IPF without COPD (n=6) by day 1, increasing to p = 0.0005 by day 22 compared to their baseline therapies, determined by changes in FVC, FEV1, PEF, and FEV1/FVC ratios. The improved FEV1/FVC ratio from 52% to 86% was clinically significant and indicated that current therapies in use are inadequate to treat patient with IPF.

The current study will expand on these findings by conducting a phase 3, double-blind placebo-controlled clinical trial to determine the effectiveness of 20mM sodium pyruvate nasal spray to decrease coughing in idiopathic pulmonary fibrosis patients. Individuals with a clinical diagnosis of idiopathic pulmonary fibrosis (as defined by the WHO and the Thoracic Society) will be solicited for participation in this phase 3 trial. Patients will have their degree of nasal inflammation and erythema, nasal cellular morphology, SaO2, and FEV1, FVC levels and blood workup recorded (baseline). Women of child-bearing age will provide a urine sample. The subjects will fill out a quality-of-life questionnaire (chronic respiratory disease questionnaire (CRDQ), and they will be given a data logbook in which they will record the number of coughs they experience each 24 hour period, for 7 days. The coughing data will be entered into the patients' logbooks and will be separated into "total coughs per 24 hours," and "night-time coughs." These data will be used to establish a baseline for coughing. After 7 days, patients will return to the clinic to begin the 21 day study where they will be given drug or placebo in a double-blinded fashion and will record their coughs daily in a logbook. Patients will return to the clinic on days 8, 15 and 22 for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a clinical diagnosis of idiopathic pulmonary fibrosis in accordance with the most recent collaborative guidelines from the American Thoracic Society, the European Respiratory Society, the Japanese Respiratory Society, and the Latin American Thoracic Association including HRCT scan and/or lung biopsy consistent with unusual interstitial pneumonia (UIP), especially honeycombing, without identifiable cause related to other ILD such as drug toxicity, occupational or environmental exposure or connective tissue disease.
* condition-related cough.
* Mild to moderate FEV1 and FVC at 50% or greater of standard
* Individuals who agree to abstain from sexual intercourse, or agree to use condoms or vaginal diaphragms or other devices designed to prevent contraception, during the entire course of the study.

Exclusion Criteria:

* Pulmonary disease other than idiopathic pulmonary fibrosis.
* Respiratory infections in the last 2 weeks.
* Clinically significant cardiac disease including uncontrolled congestive heart failure and unstable angina.
* Pregnancy (urine pregnancy test will be performed prior to enrollment).
* Females of childbearing potential age not on adequate contraception or lactating females.
* Subjects less than 18 years of age.
* Hospitalization within last 6 months due to acute exacerbation of airway disease.
* Subjects with a clinically significant abnormal chest X-ray within past 12 months.
* Medication changes within 1 month of study entry except for antiviral, antibiotic, or antimicrobial medications as well as corticosteroids, antihistamines, or anti-inflammatory medications.
* Subjects who have participated in another drug treatment study within the last month.
* Subjects with a current history of alcohol or recreational drug abuse.
* Subjects who have taken dietary supplements containing pyruvate within 24 hours prior to the screening visit.
* Subjects with metabolic diseases (diabetes, hypoglycemia, etc.).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel M Lam, MD, Principal Investigator — Family First Medical Research Center
Locations (1):
- Family First Medical Research Center, Hialeah Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wells AU. The revised ATS/ERS/JRS/ALAT diagnostic criteria for idiopathic pulmonary fibrosis (IPF)--practical implications. Respir Res. 2013;14 Suppl 1(Suppl 1):S2. doi: 10.1186/1465-9921-14-S1-S2. Epub 2013 Apr 16. PMID 23734820

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20mM Sodium Pyruvate Nasal Spray Treatment | Saline Placebo Control
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20mM Sodium Pyruvate Nasal Spray Treatment | Saline Placebo Control | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.3) | 46.5 (13.9) | 47.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 22 | 45
  Hispanic | 2 | 1 | 3
  Black | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Coughing Episodes Per Day From Baseline to Day 21.
Description: Percent change in coughing was calculated by subtracting the baseline coughs per day from the day 21 coughs per day and then dividing by the baseline coughs per day. The a priori threshold was set at a 25% or greater decrease. (An episode is defined as 5 or more coughs per hour.)
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: % change in coughing episodes
Arm/Group | 20mM Sodium Pyruvate Nasal Spray Treatment | Saline Placebo Control
Number analyzed (Participants) | 26 | 24
% change in coughing episodes | -73.2 (8.1) | -16.1 (11.0)
Statistical Analysis 1: Comparison: 20mM Sodium Pyruvate Nasal Spray Treatment vs Saline Placebo Control; Test type: Superiority; p = 0.0001, ANOVA — Sidak's test was used to adjust for multiple comparisons; Degrees of freedom, 42.19; Mean Difference (Final Values) = -57.13, 95% CI 2-sided [-63.99 to -50.27], Standard Error of Mean 2.759

2. Secondary Outcome: Percent Change in FEV1/FVC Ratios From Baseline to Day 21.
Description: The FEV1/FVC ratio was determined for baseline and day 21. The percent change was then calculated subtracting the baseline FEV1/FVC ratio from the day 21 FEV1/FVC ratio and then dividing by the baseline FEV1/FVC ratio. The a priori change was set at 12% or more.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: % change in FEV1/FVC ratios
Arm/Group | 20mM Sodium Pyruvate Nasal Spray Treatment | Saline Placebo Control
Number analyzed (Participants) | 26 | 24
% change in FEV1/FVC ratios | 27.9 (22.0) | 2.73 (5.34)
Statistical Analysis 1: Comparison: 20mM Sodium Pyruvate Nasal Spray Treatment vs Saline Placebo Control; Test type: Superiority; p < 0.0001, ANOVA; Degrees of freedom, 28.16; Mean Difference (Final Values) = 25.12, 95% CI 2-sided [13.26 to 36.99], Standard Error of Mean 4.459

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the four week study, including one week pre-study baseline.
Arm/Group | 20mM Sodium Pyruvate Nasal Spray Treatment | Saline Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 4/26 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mM Sodium Pyruvate Nasal Spray Treatment (N=26) | Saline Placebo Control (N=24)
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) — Nasal irritation lasting no more than 2 days during the first week of treatment.
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT06037408/Prot_SAP_000.pdf